CLINICAL TRIAL: NCT07279857
Title: The Impact of a Mobile Application-based Support and Counseling Program on Women's Knowledge, Attitudes and Self-efficacy in the Preconceptional Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selinay Aktaş Demir (Other)
Responsible Party: Sponsor-Investigator, Selinay Aktaş Demir, Lecturer, RN, MSc, PhD Student, Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ATLASU-AKTASDEMIR-001
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Preconception Period
Keywords: Preconception Care; Preconception Counseling; Mobile Health (mHealth); Digital Health Intervention; Women's Health; Reproductive Health; Self-Efficacy

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel groups: a mobile application-based counseling intervention group and a standard-information control group. Both groups receive their assigned intervention simultaneously, and outcomes are measured at baseline, week 4, and week 12.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment; the researcher delivering the intervention is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Women receive a four-week mobile application-based preconception counseling program including weekly modules, reminders, and messaging support.
  Interventions: Behavioral: Mobile Application-Based Preconception Counseling Program
- Control Group (Active Comparator): Women receive a standard preconception information booklet containing guideline-based educational content.
  Interventions: Behavioral: Standard Preconception Information Booklet

INTERVENTIONS:
Behavioral: Mobile Application-Based Preconception Counseling Program — A structured digital education and counseling program delivered through a mobile application, including weekly modules, reminders, and in-app messaging support.
  Arms: Intervention Group
Behavioral: Standard Preconception Information Booklet — A printed booklet providing standard guideline-based preconception information without digital follow-up.
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a mobile application-based support and counseling program on women in the preconception period. The study includes women aged 18 to 49 who plan to conceive within two years and meet the eligibility criteria. Participants are randomly assigned to an intervention group receiving structured preconception counseling through a mobile application or a control group receiving standard information via a booklet. The intervention consists of weekly educational modules delivered over four weeks, followed by follow-up assessments at 4 and 12 weeks. Primary outcomes include changes in preconception knowledge, attitudes, and self-efficacy. The study seeks to determine whether mobile health-based counseling enhances preconception preparedness compared with standard information.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of a structured mobile application-based support and counseling program designed for women in the preconception period. Preconception care plays a critical role in improving maternal and fetal outcomes by addressing biomedical, behavioral, and psychosocial risk factors before pregnancy. Despite increasing global use of mobile health technologies, there is no comprehensive mobile application-based preconception counseling program developed and evaluated in Türkiye. This study aims to address this gap by implementing a digitally delivered intervention grounded in established guidelines from the CDC and WHO.

The study includes women aged 18 to 49 who are in the preconception period, have never been pregnant, plan to conceive within two years, can use a smartphone, and have internet access. Women who are currently pregnant, health professionals, those with diagnosed psychiatric conditions, or those who have previously received preconception counseling are excluded. A total of 110 eligible participants are enrolled and randomly assigned to intervention or control groups using a simple randomization procedure generated through an online randomization system (random.org). Because the intervention requires participant engagement with content, the study is conducted as a single-blind design, with participants unaware of their group allocation.

The intervention group receives a four-week mobile application-based counseling program developed using the ADDIE (Analysis, Design, Development, Implementation, Evaluation) instructional design model. The application delivers weekly modules covering preconception care concepts, risk assessment, nutrition, supplementation, physical activity, immunization, sexually transmitted infections, environmental exposures, oral and dental health, psychosocial well-being, reproductive planning, and lifestyle behaviors such as tobacco, alcohol, and medication use. Each module includes structured educational content, reminders, and communication tools enabling researcher-participant interaction. Participants receive weekly follow-ups via messaging to identify difficulties, support adherence, and address questions. The application also includes built-in progress tracking and notification functions.

The control group receives a printed booklet containing standardized preconception information aligned with the topics covered in the intervention modules. Control group participants do not receive digital follow-up but participate in the same assessment schedule as the intervention group.

Data are collected at baseline, at week 4, and at week 12 after the start of the study. Instruments include: a descriptive information form, the Preconception Knowledge and Attitudes Scale, the General Self-Efficacy Scale, a preconception risk assessment form, and for the intervention group, the Mobile Application Usability Scale. Baseline assessments include sociodemographic characteristics, lifestyle indicators, and preconception risk factors. Week 4 assessments measure short-term changes in knowledge, attitudes, and self-efficacy. Week 12 assessments evaluate persistence of intervention effects and longer-term retention of gains.

The primary outcomes are changes in preconception knowledge, attitudes, and self-efficacy. Secondary outcomes include user-reported usability and acceptability of the mobile application. The study evaluates whether a mobile health-based digital counseling approach provides measurable benefits beyond conventional booklet-based information and whether its effects persist beyond the immediate intervention period.

The findings are expected to contribute to the development of evidence-based, scalable, digital preconception care strategies appropriate for primary health care settings, particularly in contexts where accessibility, continuity, and standardization of preconception counseling services are limited.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 49 years.
2. In the preconception period and planning to conceive within the next two years.
3. Never been pregnant.
4. Able to read and understand Turkish.
5. Having a smartphone and internet access.
6. Willing to participate and provide informed consent.

Exclusion Criteria:

1. Currently pregnant.
2. Having a diagnosed psychiatric disorder that may interfere with participation.
3. Previous participation in structured preconception counseling or training.
4. Being a health professional or a student in a health-related field.
5. Inability to use a mobile application due to cognitive, visual, or physical limitations.
6. Participation in another ongoing research study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as women are eligible to participate.
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Preconception Knowledge Score | Baseline, Week 4, Week 12
  Preconception knowledge is assessed using the Preconception Knowledge and Attitudes Scale. The primary outcome is the change in total knowledge score from baseline to week 4 and week 12. Higher scores indicate higher preconception knowledge.

SECONDARY OUTCOMES:
Change in Preconception Attitudes Score | Baseline, Week 4, Week 12
  Attitudes toward preconception health are measured using the attitude subscale of the Preconception Knowledge and Attitudes Scale. Change in attitude score is evaluated between baseline, week 4, and week 12.
Change in Self-Efficacy Score | Baseline, Week 4, Week 12
  Self-efficacy is assessed using the General Self-Efficacy Scale. The outcome measure is the change in total self-efficacy score across baseline, week 4, and week 12.
Mobile Application Usability Score | Week 4
  Usability of the mobile application is assessed using a validated usability scale. Usability is measured at week 4 among participants in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Selinay Aktaş Demir, RN, PhD Student, Principal Investigator — Atlas Üniversitesi; Ümran Oskay, PhD, Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Bayrampaşa İlçe Sağlık Müdürlüğü Aile Sağlığı Merkezleri, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No